CLINICAL TRIAL: NCT01258582
Title: Optimizing Strategies for Universal HIV Testing (The USHER Trial): Phase II
Brief Title: Two Approaches to Routine HIV Testing in a Hospital Emergency Department
Acronym: USHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rochelle Walensky, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R01 MH073445 (Phase II); R01MH073445 (NIH)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Results first posted 2012-06-05 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: HIV; Testing; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — HIV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral HIV testing (Experimental)
  Interventions: Procedure: Oral HIV screening
- Fingerstick HIV testing (Active Comparator)
  Interventions: Procedure: Fingerstick HIV screening

INTERVENTIONS:
Procedure: Oral HIV screening — Participants will undergo oral HIV screening and, if positive, further study visits for up to 6 months
  Arms: Oral HIV testing
Procedure: Fingerstick HIV screening — Participants will undergo fingerstick HIV screening and, if positive, further study visits for up to 6 months
  Arms: Fingerstick HIV testing

SUMMARY:
This study was initially designed to compare the effectiveness of two different approaches to providing routine HIV counseling, testing, and referral services in an urban hospital emergency department setting. The initial phase was closed in July 2008. The second phase of this trial consists of establishing the differences in acceptability of HIV testing based on the method of testing offered (rapid oral fluid vs. fingerstick).

DETAILED DESCRIPTION:
About 25% of HIV infected people do not know that they are infected. These people lack medical care that could prolong their lives and access to counseling services that could prevent further spread of HIV. With so many people unaware of their HIV status, there is a clear need for more readily available HIV counseling, testing, and referral services throughout the United States. The Centers for Disease Control and Prevention (CDC) recommends routine HIV testing in U.S. hospitals in which HIV infected patients make up at least 1% of the total patient population for that hospital. In the original proposal, we chose oral rapid HIV testing as we felt that this technique is noninvasive, acceptable to both patients and health care workers (without body fluid risk), and would maximize rates of HIV testing. This study directly compares acceptance rates of HIV testing as a function of the test type offered (oral vs. fingerstick) in a randomized controlled fashion.

Participants in this study will include adults who visit Brigham and Women's Hospital emergency department in Boston, Massachusetts. Participants will be randomly assigned to oral vs. fingerstick HIV testing by a designated HIV counselor and to fill out a questionnaire while waiting in the emergency room. The questionnaire will be anonymous. Participants will then be offered a rapid HIV test. Test results will be available in about 20 minutes and will be provided to participants by the HIV counselor. Participants who test positive for HIV will be offered a more definitive blood test to confirm HIV infection. The blood test results will be available 2 weeks from testing, and participants must return to the hospital to get their test results. Participants who test positive for HIV will be offered counseling support and referral services by either their assigned HIV counselor or emergency department staff member. Follow-up care appointments will also be initiated at this time. For participants who test positive for HIV, the study will last about 6 months. There will be no follow-up visits for participants who do not test positive for HIV during their emergency room visit.

ELIGIBILITY:
Inclusion Criteria:

* Waiting to receive care in the Brigham and Women's Hospital emergency room
* English- or Spanish-speaking
* Enters the emergency room when an HIV counselor is available

Exclusion Criteria:

* An estimated severity index score of 1 or 2 who have mechanical ventilation or are not deemed alert, awake, and oriented to person, place and time by the triage nurse
* HIV infected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1651 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rochelle P Walensky, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ganguli I, Collins JE, Reichmann WM, Losina E, Katz JN, Arbelaez C, Donnell-Fink LA, Walensky RP. Missed opportunities: refusal to confirm reactive rapid HIV tests in the emergency department. PLoS One. 2013;8(1):e53408. doi: 10.1371/journal.pone.0053408. Epub 2013 Jan 8. PMID 23308216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The USHER-Phase II study was conducted in the emergency department at Brigham and Women's Hospital, Boston, MA. Between May 5, 2009 and January 4, 2010, USHER-Phase II consented eligible patients for the opportunity to be offered routine opt-in, rapid HIV screening. Enrolled subjects were randomized to fingerstick or oral specimen collection.
Groups:
- Fingerstick: Fingerstick rapid HIV testing
- Oral Fluid: Oral fluid rapid HIV testing
Period: Overall Study
Arm/Group | Fingerstick | Oral Fluid
Started | 830 | 821
Completed | 548 | 563
Not Completed | 282 | 258

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingerstick | Oral Fluid | Total
Number analyzed (Participants) | 830 | 821 | 1651
Age Continuous [Mean (Standard Deviation); unit: years] | 34 (13) | 33 (13) | 33 (13)
Gender [Number; unit: participants] — Numbers in gender category do not add up to total number randomized due to missing data/numbers.
  participants
    Female | 536 | 529 | 1065
    Male | 283 | 288 | 571
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 198 | 201 | 399
  Non-Hispanic Black | 188 | 200 | 388
  Hispanic | 329 | 297 | 626
  Asian/Asain-American | 22 | 22 | 44
  Native American/Alaskan Native | 1 | 4 | 5
  Multi-racial/Other | 85 | 92 | 177
  Missing | 7 | 5 | 12
Primary Language [Number; unit: participants]
  English | 643 | 644 | 1287
  Spanish | 148 | 141 | 289
  Other | 34 | 29 | 63
  Missing | 5 | 7 | 12
Education [Number; unit: participants]
  Less than High School | 116 | 96 | 212
  High School/General Education Diploma | 255 | 261 | 516
  Some College | 198 | 222 | 420
  College Degree | 173 | 144 | 317
  Some Post-College/Graduate Degree | 67 | 82 | 149
  Missing | 21 | 16 | 37

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the HIV Test
Description: The primary outcome measure was HIV test acceptance rate defined by the proportion of participants whom accepted HIV testing among those randomized within each trial arm (fingerstick or oral fluid).
Time Frame: Assess on day subject enrolled into the study
Population: Intent to treat analysis
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Fingerstick HIV Testing: whole-blood fingerstick rapid HIV testing
- Oral HIV Testing: oral fluid rapid HIV testing
Arm/Group | Fingerstick HIV Testing | Oral HIV Testing
Number analyzed (Participants) | 830 | 821
proportion of participants | 0.67 [0.64 to 0.70] | 0.69 [0.66 to 0.72]
Statistical Analysis 1: Comparison: Fingerstick HIV Testing vs Oral HIV Testing; Sample size was chosen to detect a 10% difference in acceptance rates between two testing modality arms (90% power, 0.05 level of significance); Test type: Superiority or Other; p = 0.34, Chi-squared; The difference in the acceptance rates was estimated along with 95% confidence intervals and tested using the chi-square test; difference in the acceptance rates = -0.022, 95% CI 2-sided [-0.067 to 0.023]

ADVERSE EVENTS:
Description: The number at risk only includes subjects who consented to HIV testing after being randomized and offered a rapid HIV test.
Arm/Group | Fingerstick | Oral Fluid
Serious Adverse Events (participants affected / at risk) | 0/553 | 0/565
Other Adverse Events (participants affected / at risk) | 2/553 | 1/565
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fingerstick (N=553) | Oral Fluid (N=565)
False-positive rapid test result (Investigations) | 1 (1) | 0 (0)
Subject did not follow-up after reactive test (Investigations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes